CLINICAL TRIAL: NCT06865235
Title: Efficacy and Safety of Gonioscopy Assisted Transluminal Trabeculotomy in Patients with Primary Open-angle Glaucoma and Cataract - a Randomized Clinical Trial
Brief Title: Efficacy and Safety of Gonioscopy Assisted Transluminal Trabeculotomy in Patients with Primary Open-angle Glaucoma and Cataract.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Ciências Médicas de Minas Gerais (Other)
Collaborators: Hospital Evangélico de Belo Horizonte (Unknown)
Responsible Party: Principal Investigator, DANIEL FULGENCIO DE MOURA, Head of the Glaucoma Department, Faculdade de Ciências Médicas de Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 76604823.8.0000.5134
Record Dates: First submitted 2025-02-15; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Open Angle Glaucoma (OAG)
Keywords: Open angle glaucoma; Cataract; OAG; Goniotomy assisted transluminal trabeculotomy; GATT; trabeculotomy; Goniotomy; hemi-gatt
MeSH Terms: conditions — Glaucoma, Open-Angle; Cataract | interventions — Phacoemulsification

STUDY DESIGN:
Who Masked: Participant
Masking Description: The researcher who measures IOP
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Patients undergoing cataract surgery associated with GATT by 360º (Experimental)
  Interventions: Procedure: 360º goniotomy assisted transluminal trabeculotomy; Procedure: Phacoemulsification
- Patients undergoing cataract surgery associated with GATT by 180º (Experimental)
  Interventions: Procedure: Phacoemulsification; Procedure: 180º gonioscopy assisted transluminal trabeculotomy
- Patients undergoing only cataract surgery (Other): Control Group
  Interventions: Procedure: Phacoemulsification

INTERVENTIONS:
Procedure: 360º goniotomy assisted transluminal trabeculotomy — Open the Schlemm Canal for 360º with a polipropilen 5-0 suture via trabecular meshwork.
  Arms: Patients undergoing cataract surgery associated with GATT by 360º
Procedure: Phacoemulsification — Cataract Surgery
Procedure: 180º gonioscopy assisted transluminal trabeculotomy — Open the Schlemm Canal for 180º with a polipropilen 5-0 suture via trabecular meshwork.
  Other Names: 180º GATT; Hemi - GATT
  Arms: Patients undergoing cataract surgery associated with GATT by 180º

SUMMARY:
Prospective, randomized, , double-blind, clinical trial, comparing the variation of intraocular pressure (IOP) of patients with mild or moderate primary open-angle glaucoma (OAG) and cataract divided into three groups. All study participants should be treated for the pathology with one or more hypotensive medications or, regardless of the number of drugs, when IOP is greater than 20 mmHg and less than 26 mmHg. The two-year follow-up should also compare the reduction in the number of medications used, reoperation rate, adverse effects, visual acuity, endothelial loss, induction of astigmatism, variation in IOP according to axial diameter of the eye, anterior chamber and age, in addition to the existence of change in the quality of life of patients in the postoperative period

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 40 years or older,
* Previously included in the glaucoma departments of the participating institutions,
* Indication for cataract surgery, diagnosed by clinical examination with visual acuity (VA) equal to or worse than 20/40,
* Primary Open Angle Glaucoma (POAG), determined by the presence of typical visual field (VF) defects and/or by the aspect of the optic nerve observed at fundoscopy or retinography (increased vertical optical excavation with thinning of the neural rhyme, asymmetry of the cup/disc ratio greater than 0.2, localized loss ("notch") or defect in the retinal nerve fiber layer ("Hoyt")).
* APIC classification with amplitude greater/equal to 2 and pigmentation less than 4 on gonioscopy.
* Intraocular pressure (IOP) less than or equal to 25 mmHg before washout of hypotensive eye drops.
* IOP between 22 and 30 mmHg after washout of hypotensive eye drops or with a history of IOP greater than or equal to 21 mmHg in more than one previous care described in the medical record.

Exclusion Criteria:

Patients who have any of the following situations:

* Severe glaucoma, determined according to the Hoddap-Parrish-Anderson criteria;
* Axial diameter greater than 26 mm or less than 21.00 mm;
* Endothelial count less than 1500 cc;
* Pachymetry less than 480 or greater than 600 microns;
* Patients undergoing some type of intraocular surgery or laser procedure in the preoperative period and/or after these procedures in the postoperative period;
* Those who present some important per-operative complication during the study.
* With high risk of progression, the so-called rapid progressors, who are patients with high IOPs even with the use of many medications, regardless of the severity of the nerve injury.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Change in intraocular pressure (IOP) after surgery. | From glaucoma medications washout to 2 years after the surgery
  To evaluate the change in intraocular pressure (IOP) after surgery, in patients with mild to moderate GPAA, undergoing phacoemulsification associated with gonioscopy assisted transluminal trabeculotomy by 180º (GATT 180º) or 360º (GATT 360º), and compare the results between the groups mentioned and with similar controls, who operated only on cataracts, in a period of up to two years.
Change in the number of glaucoma medications after surgery. | From glaucoma medications washout to 2 years after the surgery
  To evaluate the change in the number of glaucoma medications applied after surgery, in patients with mild to moderate GPAA, undergoing phacoemulsification associated with gonioscopy assisted transluminal trabeculotomy by 180º (GATT 180º) or 360º (GATT 360º), and compare the results between the groups mentioned and with similar controls, who operated only on cataracts, in a period of up to two years.

SECONDARY OUTCOMES:
Prognostic factors of the surgeries. | From glaucoma medications washout to 2 years after the surgery
  Evaluate the association of IOP variation with axial eye length (AXL) in the groups.
Prognostic factors of the surgeries. | From glaucoma medications washout to 2 years after the surgery
  Evaluate the association of IOP variation with preoperative anterior chamber amplitude (ACD) in the groups.
Prognostic factors of the surgeries. | From glaucoma medications washout to 2 years after the surgery
  Evaluate the association of IOP variation with age in the groups
Survival Analysis | From glaucoma medications washout to 2 years after the surgery
  Evaluate and compare the need for new glaucoma surgeries between the groups.
Secundary changes in the eye after the surgeries | From glaucoma medications washout to 2 years after the surgery
  Evaluate the visual acuity after the surgeries and compare between them.
Secundary changes in the eye after the surgeries | From glaucoma medications washout to 2 years after the surgery
  Evaluate and compare the adverse events after the surgeries.
Secundary changes in the eye after the surgeries | From glaucoma medications washout to 2 years after the surgery
  Evaluate the decrease in corneal endothelial cell count between the groups.
Prognostic factors, and secundary changes in the eye after the surgeries | From glaucoma medications washout to 2 years after the surgery
  Evaluate and compare the change in quality of life in and between the groups.
Secundary changes in the eye after the surgeries | From glaucoma medications washout to 2 years after the surgery
  Evaluate the induction of astigmatism between the groups

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Olhos Ciências Médicas - Faculdade de Ciências Médicas de Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: Yes
all IPD collected throughout the trial
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code